CLINICAL TRIAL: NCT03226990
Title: Detection of Pressure Areas for Elastomeric Impressions With and Without Spacer Using Novel Digital Analyzing Software and Its Correlation With Retention.A Randomized Clinical Trial.
Brief Title: Detection of Pressure Areas for Two Elastomeric Impressions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nancy nader elsherbini, lecturer at faculty of oral and dental medicine,cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: prosthesis87-2017
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Free Completely Edentulous Patients
Keywords: pressure area; polyether elastomeric impression; wax spacer
MeSH Terms: interventions — Dental Impression Technique

STUDY DESIGN:
Intervention Model Description: The measurements are done on the day of denture insertion with no follow up timing intervals
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: impression technique — impression technique with and without wax spacer

SUMMARY:
Forty completely edentulous patients were selected and randomly distributed into two groups 20 patients each.Group I received complete dentures constructed from elastomeric impression with wax spacer,group II received complete dentures constructed from elastomeric impression with no wax spacer.then on time of denture insertion pressure areas were detected using pressure indicating paste and the denture retention was detected.The results showed less pressure areas in group I and more denture retention values than group II.

DETAILED DESCRIPTION:
This study was conducted to evaluate the significance of using wax spacer in the impression technique regarding the pressure areas and retention of the complete dentures constructed. Forty patients with edentulous maxillary arches were selected from the outpatient clinic of removable prosthodontics department, faculty of oral and dental medicine, Cairo university .The patients were randomly divided into two groups. Group I received dentures constructed from impression technique with wax spacer while group II received dentures constructed from impression technique with no spacer. On the day of denture insertion pressure areas were detected using pressure indicating paste and denture retention was measured using force gauge. The data was collected and analyzed using student's t-test.

ELIGIBILITY:
Inclusion Criteria:

- completely edentulous upper and lower arches. well to moderately developed ridges saliva of average viscosity and amount with normal temporomandibular joint

Exclusion Criteria:

diabetic patients radiation therapy signs of inflammation, ulceration or hyperplasia neurological disorders clicking or mandibular deviation.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
pressure areas | 1month
  pressure indicating paste on the fitting surface ,then the surface was captured then saved as JPEG format then Analysis was done using Image J software

SECONDARY OUTCOMES:
denture retention | 1 month
  using force gauge to give retentive values in Newtons

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Nader Elsherbini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masri R, Driscoll CF, Burkhardt J, Von Fraunhofer A, Romberg E. Pressure generated on a simulated oral analog by impression materials in custom trays of different designs. J Prosthodont. 2002 Sep;11(3):155-60. PMID 12237795
- [Background] Wang CW, Shao Q, Sun HQ, Mao MY, Zhang XW, Gong Q, Xiao GN. Influence of inner circular sealing area impression method on the retention of complete dentures. Braz Dent J. 2015 Mar-Apr;26(2):198-202. doi: 10.1590/0103-6440201300383. Epub 2015 Apr 1. PMID 25831114
- [Background] Al-Ahmar AO, Lynch CD, Locke M, Youngson CC. Quality of master impressions and related materials for fabrication of complete dentures in the UK. J Oral Rehabil. 2008 Feb;35(2):111-5. doi: 10.1111/j.1365-2842.2007.01796.x. Epub 2007 Dec 5. PMID 18053059